CLINICAL TRIAL: NCT02007213
Title: Development of a Proxy Motor Outcome Measure in Young Children With Neuromuscular Disease
Status: Terminated | Type: Observational
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140023; 14-NR-0023
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-05-06

CONDITIONS: Neuromuscular Disease
Keywords: Neuromuscular Disease; Motor Function; Proxy Reported Outcome; Young Children
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Patient reported outcomes (PROs) instruments are often used to measure meaningful treatment benefit or risk in clinical trials. PROs allow patients voices to be heard in ways that assist healthcare clinicians to address treatment effects and individual patient preferences. Unfortunately, infants and young children, especially those with a debilitating disease, such as neuromuscular disorders (NMD), may be less able to provide clear and concise information about treatment effects. In this case, we often defer to parents and guardians (to be referred to collectively as parents throughout protocol) to provide their perception of their child s overall health and wellbeing. Including parents in the assessment process recognizes the unique knowledge parents have of their child s development, reinforces their central role in implementing interventions, and aids in their ability to make better-informed healthcare decisions [1]. Yet, most parent-reports for young children are confined to overall quality of life (QoL). While QoL is an important area of assessment, its meaning varies among different ages and populations, and its results are often not precise enough to reveal small differences within samples [2]. A more specific area of concern in children with NMD is early-onset muscle weakness leading to difficulties in motor function.

The current lack of patient-centered, sensitive measures (based on motor function and item difficulty hierarchy) that are suited for repeated assessments in infants and young children with NMD represents a major obstacle to the rapid translation of promising therapeutic interventions from preclinical models to clinical research studies. Multiple clinical outcome measures used at a single time-point for capturing a child s functional status are burdensome, difficult to interpret and do not provide us with comprehensive, meaningful information to detect changes following an intervention [3]. Psychometric measures that can be completed by parents make it possible to collect a considerable amount of data over many time-points rather than being limited to a single clinical observation. Moreover, a parent-observational measure that focuses on their child s functional performance in their real-life will maximize the ecological validity of measures of motor development used for clinical trials.

Objective: To develop a parent reported observational measure of motor development in infants and young children, which will serve as a complimentary tool to clinical observation by reporting motor function as observed in the home setting and which will be used in clinical trials.

Study population: Parents of children aged 0-5 with neuromuscular disease and neuromuscular experts in pediatrics.

Design: Qualitative (parent interviews, focus groups) and quantitative study (analysis of newly developed questionnaire)

Outcome Measures: parental responses to phone interviews, neuromuscular expert responses to focus groups, parental responses to cognitive interviews, validity and reliability of newly developed questionnaire

DETAILED DESCRIPTION:
Patient reported outcomes (PROs) instruments are often used to measure meaningful treatment benefit or risk in clinical trials. PROs allow patients voices to be heard in ways that assist healthcare clinicians to address treatment effects and individual patient preferences. Unfortunately, infants and young children, especially those with a debilitating disease, such as neuromuscular disorders (NMD), may be less able to provide clear and concise information about treatment effects. In this case, we often defer to parents and guardians (to be referred to collectively as parents throughout protocol) to provide their perception of their child s overall health and wellbeing. Including parents in the assessment process recognizes the unique knowledge parents have of their child s development, reinforces their central role in implementing interventions, and aids in their ability to make better-informed healthcare decisions [1]. Yet, most parent-reports for young children are confined to overall quality of life (QoL). While QoL is an important area of assessment, its meaning varies among different ages and populations, and its results are often not precise enough to reveal small differences within samples [2]. A more specific area of concern in children with NMD is early-onset muscle weakness leading to difficulties in motor function.

The current lack of patient-centered, sensitive measures (based on motor function and item difficulty hierarchy) that are suited for repeated assessments in infants and young children with NMD represents a major obstacle to the rapid translation of promising therapeutic interventions from preclinical models to clinical research studies. Multiple clinical outcome measures used at a single time-point for capturing a child s functional status are burdensome, difficult to interpret and do not provide us with comprehensive, meaningful information to detect changes following an intervention [3]. Psychometric measures that can be completed by parents make it possible to collect a considerable amount of data over many time-points rather than being limited to a single clinical observation. Moreover, a parent-observational measure that focuses on their child s functional performance in their real-life will maximize the ecological validity of measures of motor development used for clinical trials.

Objective: To develop a parent reported observational measure of motor development in infants and young children, which will serve as a complimentary tool to clinical observation by reporting motor function as observed in the home setting and which will be used in clinical trials.

Study population: Parents of children aged 0-5 with neuromuscular disease and neuromuscular experts in pediatrics.

Design: Qualitative (parent interviews, focus groups) and quantitative study (analysis of newly developed questionnaire)

Outcome Measures: parental responses to phone interviews, neuromuscular expert responses to focus groups, parental responses to cognitive interviews, validity and reliability of newly developed questionnaire

ELIGIBILITY:
* INCLUSION CRITERIA
* Parent or guardian who has primary responsibility for care (hereafter referred to as parent ) of an infant or child(ren) under the age of 6 years who has been diagnosed with an early onset neuromuscular disorder confirmed by muscle biopsy and/or DNA testing. Medical records documenting the muscle biopsy and/or genetic testing will be submitted to the investigators.
* Ability to provide consent
* Age 18 years and above
* Sufficient English language skills to read and participate in discussions about the study questionnaire
* For the focus group of experts:

Expertise (at least 5 years experience in pediatric neuromuscular disease or questionnaire development). Experts will representatives from the following categories:

* pediatric therapists (physical, occupational, speech, respiratory therapists)
* pediatric medical doctors
* nurses and nurse practitioners
* social scientists with expertise in questionnaire development
* patient advocacy group representatives

EXCLUSION CRITERIA

-Participants with a reported history of emotional distress when discussing their child s illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-12-05; Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Parental responses to phone interviews, neuromuscular expert responses to focus groups, parental responses to cognitive interviews, validity and reliability of newly developed questionnaire. | 2-4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Katherine G Meilleur, C.R.N.P., Principal Investigator — National Institute of Nursing Research (NINR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Skellern CY, Rogers Y, O'Callaghan MJ. A parent-completed developmental questionnaire: follow up of ex-premature infants. J Paediatr Child Health. 2001 Apr;37(2):125-9. doi: 10.1046/j.1440-1754.2001.00604.x. PMID 11328465
- [Background] DeWalt DA, Rothrock N, Yount S, Stone AA; PROMIS Cooperative Group. Evaluation of item candidates: the PROMIS qualitative item review. Med Care. 2007 May;45(5 Suppl 1):S12-21. doi: 10.1097/01.mlr.0000254567.79743.e2. PMID 17443114
- [Background] Tucker CA, Gorton GE, Watson K, Fragala-Pinkham MA, Dumas HM, Montpetit K, Bilodeau N, Ni P, Hambleton RK, Haley SM. Development of a parent-report computer-adaptive test to assess physical functioning in children with cerebral palsy I: lower-extremity and mobility skills. Dev Med Child Neurol. 2009 Sep;51(9):717-24. doi: 10.1111/j.1469-8749.2009.03266.x. Epub 2009 May 27. PMID 19486108